CLINICAL TRIAL: NCT05848817
Title: Patient Reported Satisfaction With Contoura LASIK Utilizing the Phorcides Analytic Software
Status: Completed | Type: Observational
Sponsor: Mann Eye Institute (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: PB-23-01
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Contoura LASIK: Subjects receiving Phorcides Planned Contoura LASIK.
  Interventions: Device: Contoura LASIK

INTERVENTIONS:
Device: Contoura LASIK — Subjects receiving Phorcides Planned Contoura LASIK

SUMMARY:
The objective is to determine the percentage of subjects satisfied (Completely Satisfied or Very Satisfied) with vision after Phorcides Planned Contoura LASIK.

DETAILED DESCRIPTION:
This study is a single site, single-arm, prospective, observational study of subject satisfaction, after successful bilateral LASIK surgery. Subjects will be assessed pre-operatively, operatively and at 1 week, 1 month, and 3 months post-operatively. Clinical evaluations will include measurement of visual acuity, manifest refraction, and topography, aberrometry, and administration of the OSDI and PROWL questionnaires.

ELIGIBILITY:
Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Appropriate candidate for uncomplicated bilateral LASIK surgery
* Gender: Males and Females.
* Age: 21 to 39 years of age.
* Refractive error range - SE refractive errors up to 0.00 to -9.00 D with maximum cylinder up to 3.00 D and sphere ≤ -8.00 D.
* If currently wearing contact lenses:

  * Soft CTL wearers discontinue for minimum 3 days
  * RGP CTL wearers discontinue for 1 month per decade of wear
  * Stable refraction (2 consecutive manifest refractions within 0.25 SE)
  * Stable K readings (2 consecutive K readings in 2 consecutive visits)
* Residual bed thickness 250um or greater
* Willing and able to comply with scheduled visits and other study procedures.
* Pre-surgery BCDVA of 20/20 (0.00 logMAR) or better in each eye.

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Subjects with history of previous ocular surgery.
* Subjects with topographic evidence of keratoconus, or ectasia.
* Subjects with autoimmune diseases.
* Subjects who are pregnant or nursing.
* Systemic disease likely to affect wound healing, such as diabetes and severe atopy.
* Any ocular disease (including un-controlled dry eye) which in the investigator's opinion would affect the outcome of refractive surgery.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Ages: 21 Years to 39 Years | Sex: All
Age Groups: Adult
Study Population: Subjects 21 to 39 years of who are appropriate candidates for laser refractive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Brunson, OD, Principal Investigator — Mann Eye Institute
Locations (1):
- Mann Eye Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Contoura LASIK
Started | 50; 100 eyes
Completed | 50; 100 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Arm/Group | Contoura LASIK
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subject Satisfaction
Description: Percentage of subjects satisfied with vision after Phorcides Planned Contoura LASIK (answering Completely Satisfied or Very Satisfied on PROWL Questionnaire Question #1.
Time Frame: 3 Months Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Contoura LASIK
Number analyzed (Participants) | 50
Participants | 50

2. Secondary Outcome: Number of Eyes With Post-op Spherical Equivalent Within +/- 0.50 D
Time Frame: 3 Months Postoperative
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Contoura LASIK
Number analyzed (Participants) | 50
Number analyzed (eyes) | 100
eyes | 90

3. Other Pre Specified Outcome: PROWL Questionnaire
Description: PROWL-SS can be used to assess satisfaction with vision and the existence, bothersomeness and impact on usual activities in the last 7 days of four visual symptoms - double images (8 items), glare (8 items), halos (8 items) and starbursts (8 items). Subjects select one of 6 responses for each question. Responses are scaled from 0 to 100, with 0 being a worse overall outcome and 100 being a better overall outcome for the existence, bothersomeness and impact on usual activities in the last 7 days of four visual symptoms - double images (8 items), glare (8 items), halos (8 items) and starbursts (8 items).
Time Frame: 3 Months Postoperative
Measure: Mean (Standard Deviation); unit: score on a scale (0 to 100)
Arm/Group | Contoura LASIK
Number analyzed (Participants) | 50
score on a scale (0 to 100)
  Satisfaction score | 94.8 (8.9)
  Double image score | 99.4 (4.6)
  Glare score | 97.7 (5.9)
  Halo Score | 94.2 (7.4)
  Starburst score | 93.3 (8.8)

4. Other Pre Specified Outcome: OSDI Score
Description: The OSDI© is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease. The OSDI© is a valid and reliable instrument for measuring dry eye disease (normal, mild to moderate, and severe) and effect on vision-related function.
Time Frame: 3 Months Postoperative
Measure: Mean (Standard Deviation); unit: score on a scale (0 to 100)
Arm/Group | Contoura LASIK
Number analyzed (Participants) | 50
score on a scale (0 to 100) | 7.5 (6.7)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Contoura LASIK
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT05848817/Prot_SAP_000.pdf